CLINICAL TRIAL: NCT04682301
Title: Tailoring Shared Decision Making for Lung Cancer Screening in Persons With HIV (PWH)
Brief Title: Tailoring Shared Decision Making for Lung Cancer Screening in Persons Living With HIV
Status: Completed | Type: Observational
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Matthew Triplette, Associate Professor, Fred Hutchinson Cancer Center
Other Study IDs: RG1121165; NCI-2020-08393 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10557 (Other: Fred Hutch/University of Washington Cancer Consortium); P30CA015704 (NIH)
Record Dates: First submitted 2020-12-09; First posted 2020-12-23 (Actual); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Behavior Therapy; Focus Groups; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Aims I-II: AIM I: Participants attend a focus group over 1-1.5 hours providing feedback on refining potential methods of SDM.
  AIM II: Participants receive the SDM intervention developed in Aim I and provide feedback. Participants may attend a telephone interview over 45 minutes 1 month later.
  Interventions: Behavioral: Behavioral Intervention; Other: Discussion (focus group); Other: Discussion (feedback on SDM); Other: Interview; Other: Survey Administration

INTERVENTIONS:
Behavioral: Behavioral Intervention — Receive SDM intervention
  Other Names: Behavior Conditioning Therapy; Behavior Modification; Behavior or Life Style Modifications; Behavior Therapy; Behavioral Interventions; Behavioral Modification; Behavioral Therapy; Behavioral Treatment; Behavioral Treatments
Other: Discussion (focus group) — Attend focus group
  Other Names: Discuss
Other: Discussion (feedback on SDM) — Provide feedback on SDM
  Other Names: Discuss
Other: Interview — Attend a telephone interview
Other: Survey Administration — Ancillary studies

SUMMARY:
This study tailors a shared decision making intervention for lung cancer screening in persons living with human immunodeficiency virus (HIV). Information collected in this study may help doctors better understand how to perform lung cancer screening in persons living with HIV, so as to enhance shared decision making in persons living with HIV.

DETAILED DESCRIPTION:
OUTLINE:

AIM I: Participants attend a focus group over 1-1.5 hours providing feedback on refining potential methods of shared decision making (SDM).

AIM II: Participants receive the SDM intervention developed in Aim I and provide feedback. Participants may attend a telephone interview over 45 minutes 1 month later.

ELIGIBILITY:
Inclusion Criteria:

* AIM I: Patients with human immunodeficiency virus (PWH) enrolled in the local UW HIV cohort and primary providers at Madison Clinic and other Seattle-based clinics serving PWH
* AIM I: Using proposed United States Preventive Services Task Force (USPSTF) guidelines, participants enrolled in the registry who are current or former smokers, report >= 20 pack-years smoking history, and >= 50 years old (n=165) will be eligible for recruitment
* AIM I: Clinicians (medical doctors, physicians assistants and nurse practitioners) who provide primary care for PWH (n=48) will be eligible
* AIM II: PWH who are eligible for lung cancer screening (LCS) based on proposed USPSTF criteria

Exclusion Criteria:

* Those found to be ineligible for LCS on coordinator review
* Are non-English speaking or have cognitive dysfunction that would prevent participation in SDM

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: PWH enrolled in the local University of Washington (UW) HIV cohort and primary providers at Madison Clinic
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2021-02-05 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Triplette, MD, MPH, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Murphy NR, Crothers K, Snidarich M, Budak JZ, Brown MC, Weiner BJ, Giustini N, Caverly T, Durette K, DeCell K, Triplette M. The Use of a Tailored Decision Aid to Improve Understanding of Lung Cancer Screening in People With HIV. Chest. 2025 Jan;167(1):259-269. doi: 10.1016/j.chest.2024.07.147. Epub 2024 Jul 29. PMID 39084517

RESULTS

PARTICIPANT FLOW:
Groups:
- Observational: AIM I: Participants attend a focus group over 1-1.5 hours providing feedback on refining potential methods of SDM.
  AIM II: Participants receive the SDM intervention developed in Aim I and provide feedback. Participants may attend a telephone interview over 45 minutes 1 month later.
  Behavioral Intervention: Receive SDM intervention
  Discussion (focus group): Attend focus group
  Discussion (feedback on SDM): Provide feedback on SDM
  Interview: Attend a telephone interview
  Survey Administration: Ancillary studies
Period: Overall Study
Arm/Group | Observational
Started (Includes participants in focus groups only (Aim I), the shared decision making only (Aim II), and those enrolled in both Aim I and Aim II.) | 102
Completed (Includes only individuals who participated in Aim II (100% completion of individuals enrolled in Aim II).) | 40
Not Completed | 62
Not completed — Participant enrolled in Aim I only. | 60
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Groups:
- Aims I-II: AIM I: Participants attend a focus group over 1-1.5 hours providing feedback on refining potential methods of SDM.
  AIM II: Participants receive the SDM intervention developed in Aim I and provide feedback. Participants may attend a telephone interview over 45 minutes 1 month later.
  Behavioral Intervention: Receive SDM intervention
  Discussion (focus group): Attend focus group
  Discussion (feedback on SDM): Provide feedback on SDM
  Interview: Attend a telephone interview
  Survey Administration: Ancillary studies
Arm/Group | Aims I-II
Number analyzed (Participants) | 102
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 58.5 [55 to 63]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 82
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 74
  Race: Black or African American | 9
  Race: American Indian or Alaska Native | 1
  Race: Asian | 4
  Race: Native Hawaiian or Pacific Islander | 0
  Race: More than one race | 9
  Race: Other race -- described as Hispanic or Latinx | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 102

OUTCOME MEASURES:

1. Primary Outcome: Focus Group Analysis (Aim I)
Description: All focus groups will be recorded and transcribed. Will use a framework analysis approach which combines both inductive and deductive methods where generated themes are mapped onto an implementation framework, specifically the Tailored Implementation of Chronic Diseases (TICD) checklist. Codes will then be analyzed through a constant comparison method to determine key themes. Will analyze all focus groups in real time to make iterative changes to the focus group guide based on feedback and refining potential methods of shared decision making (SDM). Pre-/post-SDM survey data will be collected via tablet, with a paper option if desired.
  Effectively, number of participants who complete focus group participation for analysis.
Time Frame: During focus participation, an average of 1-1.5 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Aims I-II
Number analyzed (Participants) | 102
Participants | 43

2. Primary Outcome: Improvement in Lung Cancer Screening Knowledge (LKS), According to Pre- vs. Post-intervention Scores (Aim II)
Description: The primary outcome was change in knowledge of LCS after using the tailored decision aid. We used two validated measures of LCS knowledge, the LCS-12 and LKS-7, to evaluate knowledge of risks, benefits, and characteristics of LCS. The LCS-12 includes twelve multiple-choice questions which assess knowledge of lung cancer risk, characteristics of LCS, and benefits and harms of LCS. The LKS-7 uses seven questions assessing understanding of the harms and benefits LCS, incidental findings, and the screening process. Our enrollment target was 40-50 patients to achieve greater than 90% power to observe a difference similar to a prior study in pre- and post-SDM knowledge of screening harms (69% to 93%). Minimum score of 0 for LCS-12 and LKS-7, indicating no improvement from pre- to post-intervention assessment on LCS knowledge; maximum score of 12 for LCS-12 and 7 for LKS-7. Higher score represents better outcome, or greater improvement from pre- to post-intervention on measures of LKS.
Time Frame: During shared decision-making participation, an average of 1 hour
Population: Includes subset of individuals who completed shared decision-making visit in interventional Aim only.
Measure: Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Aims I-II
Number analyzed (Participants) | 40
score on a scale
  LCS-12 | 2.8 [2.1 to 3.5]
  LKS-7 | 1.1 [0.6 to 1.6]

3. Primary Outcome: Decision of Cancer Screening (DCS) (Aim II)
Description: The Decision of cancer screening (DCS) was used to evaluate participants' decisional conflict after SDM visits. The ten-item lower literacy DCS was selected with possible scores ranging from 0 (minimum; no decisional conflict) to 100 (maximum; extremely high decisional conflict), with possible sub-scores for resulting feelings of uncertainty, feeling informed, clarity of values regarding risks and benefits, and feeling supported. Each question has options for yes (0), unsure (2), and no (4); answers are summed, divided by ten, then multiplied by 25 to provide the overall DCS. Lower scores represent a better outcome, or no/low decisional conflict.
Time Frame: During shared decision-making participation, an average of 1 hour
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Aims I-II
Number analyzed (Participants) | 40
score on a scale | 0 [0 to 5]

4. Primary Outcome: Acceptability of Intervention Measure (AIM) (Aim II)
Description: The AIM was used to evaluate the acceptability of the intervention for participants. The AIM is a four-item measure to assess the acceptability of a given intervention, in this case the decision aid, producing responses on a scale from 1 (completely disagree) to 5 (completely agree) and higher scores indicating greater acceptability.
  The score is calculated by taking the mean of the four responses. Scores range from 1-5.
Time Frame: During shared decision-making participation, an average of 1 hour
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Aims I-II
Number analyzed (Participants) | 40
score on a scale | 4.1 [4 to 5]

5. Primary Outcome: Fidelity (Aim II)
Description: Fidelity summarized as median percent of a 10-item checklist completed. Higher percentages represented a better outcome, or greater fidelity to the intervention/completion of items throughout intervention. Minimum percentage of completion is 0; maximum percentage of completion is 100.
Time Frame: During shared decision-making participation, an average of 1 hour
Measure: Median (Inter-Quartile Range); unit: percentage of completion
Arm/Group | Aims I-II
Number analyzed (Participants) | 40
percentage of completion | 100 [97.5 to 100]

ADVERSE EVENTS:
Time Frame: Up to 1.5 years after participant enrollment.
Description: Definition of adverse and serious adverse event do not vary from clinicaltrials.gov definition.
Arm/Group | Aims I-II
All-Cause Mortality (participants affected / at risk) | 3/102
Serious Adverse Events (participants affected / at risk) | 0/102
Other Adverse Events (participants affected / at risk) | 0/102

LIMITATIONS AND CAVEATS:
Limitations of this study are largely related to this being a pilot single-center study with no control arm. Additionally, it was implemented in a clinic already familiar with having regular SDM conversations regarding LCS which may limit generalizability to a primary care setting. Our study did not assess the durability of this improvement over weeks to months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/01/NCT04682301/Prot_SAP_000.pdf